CLINICAL TRIAL: NCT02940574
Title: Oxytocin-based Pharmacotherapy for Autism Spectrum Disorders: Investigating the Neural and Behavioral Effects of a Promising Intervention Approach
Brief Title: Neural and Behavioral Effects of Oxytocin in Autism Spectrum Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: The Branco Weiss Fellowship (Other); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Kaat Alaerts, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S56327; 2014-000586-45 (EudraCT Number)
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Results first posted 2020-02-13 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Autism Spectrum Disorders
Keywords: Oxytocin; Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Syntocinon (Oxytocin, product code RVG 03716) (Experimental): Administration via nasal spray
  Interventions: Drug: Syntocinon (Oxytocin)
- Placebo (Physiological water(sodium chloride (NaCl) solution)) (Placebo Comparator): Administration via nasal spray
  Interventions: Other: Placebo (Physiological water (solution of sodium chloride (NaCl) in water))

INTERVENTIONS:
Drug: Syntocinon (Oxytocin) — Syntocinon nasal spray. A single dose (24IU) of nasal spray (3 puffs of 4IU per nostril), followed by 4 weeks of a daily single dose (24IU; 3 puffs of 4IU per nostril) of nasal spray
  Arms: Syntocinon (Oxytocin, product code RVG 03716)
Other: Placebo (Physiological water (solution of sodium chloride (NaCl) in water)) — Placebo nasal spray. A single dose (24IU) of nasal spray (3 puffs of 4IU per nostril), followed by 4 weeks of a daily single dose (24IU; 3 puffs of 4IU per nostril) of nasal spray
  Arms: Placebo (Physiological water(sodium chloride (NaCl) solution))

SUMMARY:
The current trial aims to explore the neural and behavioral effects of oxytocin in autism spectrum disorders (ASD). Oxytocin is a nonapeptide produced by the paraventricular and supraoptic nuclei of the hypothalamus and is known to play a pivotal role in a variety of complex social behaviors. Initial studies showed that intranasal administration of oxytocin can have a positive effect on social functioning in ASD.

However, future studies are necessary to explore whether and how oxytocin effects neural processes in the brain underlying these behavioral improvements. This trial will not only measure behavioral enhancements, but will specifically focus on elucidating the associated neurophysiological changes by guiding the administration of oxytocin with regular neurophysiological assessments.

DETAILED DESCRIPTION:
The present study is a monocentric, between-subjects, randomized, placebo-controlled trial. The investigators will recruit approximately 40 young-adult, male individuals with a clinical diagnosis of Autism Spectrum Disorder (ASD). Participants will be randomly allocated to an experimental group (Oxytocin (OT)) and a control group (Placebo (PL)). All participants will receive the same frequency and duration of intervention. Behavioral and neural outcome measures will be assessed at multiple time points in a period of a year. Participants will be tested at 5 occasions: before and after a single dose of nasal spray, after multiple doses of nasal spray (1 daily dose of nasal spray during 4 weeks), after a 4-week retention period and after a 1-year retention period. At each time point participants will be tested at both the behavioral and neural level. Test performance of both participant groups (OT vs PL) will be compared by measuring reaction times and accuracy rates in a computerized task assessing a person's ability to recognize bodily emotional states from point light displays. In addition, attachment, social functioning, restricted behaviour, general quality of life and mood will be assessed via self-reported questionnaires.

Functional MRI measurements will be performed in a 3T MR Philips Intera scanner. Before scanning, subjects will undergo a training session to familiarize them with the task instructions. In addition to the fMRI measurements, resting state fMRI and Diffusion Tensor Imaging (DTI) will also be performed to reveal alterations of the functional and structural connectivity between critical regions.

Statistical analysis of the behavioral data will have a between-subject factor of group (OT vs PL) and within-subject factors of time (change-from-baseline). Image analysis will be performed with Statistical Parametric Mapping (SPM) software. The investigators will contrast for either decreased or increased activation, as different regions may show divergent changes due to the received nasal spray (either OT or PL).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Autism Spectrum Disorder, Asperger Syndrome or Autism
* Male
* Age between 18 and 40 years old

Exclusion Criteria:

* Associated neuro(psycho)logical disorder (i.e. epilepsy, concussion, stroke)
* Eye sight worse than + or - 7
* Genetic syndrome
* Color blindness
* Any contraindication to neuroimaging research as assessed with the MRI screening list:

MRI contraindications:

pacemaker, implanted defibrillator, ear implant / a cochlear implant, insulin or implanted pump, a neurostimulator or VP shunt, any metallic object in the eyes (metallic fragments)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Alaerts, PhD, Principal Investigator — KU Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were mainly recruited from the Expertise Centrum Autisme of the UZ Leuven between April 2015 and December 2016. Recruitment and patient contact were facilitated by our collaboration with Prof. Dr. Jean Steyaert, head of UZ Leuven ECA.
Period: From Study Start to 1-month Follow-up
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Started | 22 | 18
Completed | 21 (Discontinued intervention (N=1): self-termination unrelated to treatment) | 18 (All participants completed, but data from 1 participant was not included in analyses.)
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: 1-year Follow-up
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Started | 21 | 18
Completed | 18 | 14
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution)) | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Assessed via self-report.
  years | 25.00 (4.86) | 24.00 (5.55) | 24.38 (5.11)
Sex: Female, Male [Count of Participants; unit: Participants] — Only men were included in the study.
  Participants
    Female | 0 | 0 | 0
    Male | 22 | 18 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 18 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 22 | 18 | 38
Total IQ [Mean (Standard Deviation); unit: units on a scale] — 6-subtest short version of the Wechsler Adult Intelligence Scale-IV Dutch version: Block design, Digit span, Similarities, Vocabulary, Symbol search and Visual puzzles
  units on a scale | 102.27 (12.45) | 104.61 (21.59) | 104.24 (15.72)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Brain Activity During Task (Task-based fMRI) After a Single Dose of Nasal Spray
Description: Change From Baseline in Task-related Brain Activity During Biological Motion Recognition Task (Task-based fMRI) After a Single Dose of Nasal Spray BOLD response (Blood-oxygen-level-dependent response)
Time Frame: Value at 30 minutes minus value at baseline
Population: 1 subject lost in Syntocinon group due to subject withdrawal.
  1 subject lost in Placebo group due to low data quality (excessive in-scanner head motion)
Measure: Mean (Standard Deviation); unit: Change-from-baseline (BOLD response)
Groups:
- Syntocinon (Oxytocin, Product Code RVG 03716): Administration via nasal spray
  Syntocinon (Oxytocin): Syntocinon nasal spray. A single dose (24IU) of nasal spray (3 puffs of 4IU per nostril).
- Placebo (Physiological Water(Sodium Chloride (NaCl) Solution)): Administration via nasal spray
  Placebo (Physiological water (solution of sodium chloride (NaCl) in water)): Placebo nasal spray.
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 21 | 17
Change-from-baseline (BOLD response)
  Brain activity - Superior temporal sulcus | 0.11 (0.49) | -0.26 (0.72)
  Brain activity - Amygdala | -0.15 (0.50) | -0.16 (0.58)

2. Primary Outcome: Change From Baseline in Brain Activity During Task (Task-based fMRI) After 4 Weeks of Nasal Spray
Description: Change From Baseline in Task-related Brain Activity During Biological Motion Recognition Task (Task-based fMRI) after 4 weeks of nasal spray BOLD response (Blood-oxygen-level-dependent response)
Time Frame: Value at 4 weeks minus value at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change-from-baseline (BOLD response)
Groups:
- Syntocinon (Oxytocin, Product Code RVG 03716): Administration via nasal spray
  Syntocinon (Oxytocin): Syntocinon nasal spray. 4 weeks of a daily single dose (24IU; 3 puffs of 4IU per nostril) of nasal spray
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 21 | 17
Change-from-baseline (BOLD response)
  Brain activity - Superior temporal sulcus | -0.10 (0.59) | -0.29 (0.68)
  Brain activity - Amygdala | -0.09 (0.46) | 0.06 (0.45)

3. Primary Outcome: Change From Baseline in Brain Activity During Task (Task-based fMRI) After 8 Weeks, Including 4 Weeks Without Nasal Spray
Description: Change From Baseline in Task-related Brain Activity During Biological Motion Recognition Task (Task-based fMRI) after 8 weeks, including 4 weeks without nasal spray BOLD response (Blood-oxygen-level-dependent response)
Time Frame: Value at 8 weeks minus value at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change-from-baseline (BOLD response)
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 21 | 17
Change-from-baseline (BOLD response)
  Brain activity - Superior temporal sulcus | -0.21 (0.58) | -0.16 (0.66)
  Brain activity - Amygdala | -0.18 (0.52) | 0.04 (0.56)

4. Primary Outcome: Change From Baseline in Brain Activity During Task (Task-based fMRI) After 52 Weeks, Including 48 Weeks Without Nasal Spray
Description: Change From Baseline in Task-related Brain Activity During Biological Motion Recognition Task (Task-based fMRI) after 52 weeks, including 48 weeks without nasal spray BOLD response (Blood-oxygen-level-dependent response)
Time Frame: Value at 52 weeks minus value at baseline
Population: 1 subject lost in Syntocinon group due to subject withdrawal. (+ 3 additional participants lost for 1-year follow-up)
  1 subject lost in Placebo group due to low data quality (excessive in-scanner head motion) (+ 3 additional participants lost for 1-year follow-up)
Measure: Mean (Standard Deviation); unit: Change-from-baseline (BOLD response)
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 18 | 14
Change-from-baseline (BOLD response)
  Brain activity - Superior temporal sulcus | -0.18 (0.56) | -0.48 (0.73)
  Brain activity - Amygdala | -0.21 (0.51) | 0.03 (0.40)

5. Primary Outcome: Change From Baseline in Brain Connectivity During Rest (Resting-state fMRI) After a Single Dose of Nasal Spray
Description: Change From Baseline in Brain Connectivity During Rest (Resting-state fMRI) After a Single Dose of Nasal Spray
  Amygdala connectivity (Change-from-baseline z-transformed r-value) Higher z-transformed r-value indicates higher connectivity (higher correlated brain activity)
Time Frame: Value at 30 minutes minus value at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change-from-base z-transformed r-value
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 21 | 17
Change-from-base z-transformed r-value | -0.07 (0.21) | 0.03 (0.20)
Statistical Analysis 1: Comparison: Syntocinon (Oxytocin, Product Code RVG 03716) vs Placebo (Physiological Water(Sodium Chloride (NaCl) Solution)); Test type: Other — Linear mixed-effect analyses, exploring whether a single-dose of OT could reduce amygdala connectivity, revealed a tentative effect of 'treatment' (F(1,36)=2.00; p=.08 (one-sided)); p < 0.08, Mixed Models Analysis — Linear mixed-effect analyses, exploring whether a single-dose of OT could reduce amygdala connectivity, revealed a tentative effect of 'treatment' (F(1,36)=2.00; p=.08 (one-sided)); (F(1,36)=2.00; p=.08 (one-sided))

6. Primary Outcome: Change From Baseline in Brain Connectivity During Rest (Resting-state fMRI) After 4 Weeks of Nasal Spray
Description: Change from baseline in brain connectivity during rest (resting-state fMRI) after 4 weeks of nasal spray
  Amygdala connectivity (Change-from-baseline z-transformed r-value) Higher z-transformed r-value indicates higher connectivity (higher correlated brain activity)
Time Frame: Value at 4 weeks minus value at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change-from-base z-transformed r-value
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 21 | 17
Change-from-base z-transformed r-value | -0.04 (0.22) | 0.11 (0.21)

7. Primary Outcome: Change From Baseline in Brain Connectivity During Rest (Resting-state fMRI) After 8 Weeks, Including 4 Weeks Without Nasal Spray
Description: Change from baseline in brain connectivity during rest (resting-state fMRI) after 8 weeks, including 4 weeks without nasal spray
  Amygdala connectivity (Change-from-baseline z-transformed r-value) Higher z-transformed r-value indicates higher connectivity (higher correlated brain activity)
Time Frame: Value at 8 weeks minus value at baseline
Measure: Mean (Standard Deviation); unit: Change-from-base z-transformed r-value
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 21 | 17
Change-from-base z-transformed r-value | -0.07 (0.17) | 0.13 (0.18)

8. Primary Outcome: Change From Baseline in Brain Connectivity During Rest (Resting-state fMRI) After 52 Weeks, Including 48 Weeks Without Nasal Spray
Description: Change from baseline in brain connectivity during rest (resting-state fMRI) after 52 weeks, including 48 weeks without nasal spray
  Amygdala connectivity (Change-from-baseline z-transformed r-value) Higher z-transformed r-value indicates higher connectivity (higher correlated brain activity)
Time Frame: Value at 52 weeks minus value at baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Change-from-base z-transformed r-value
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 18 | 14
Change-from-base z-transformed r-value | -0.06 (0.20) | 0.11 (0.23)

9. Secondary Outcome: Change From Baseline in Performance on the Emotion Recognition Task (Accuracy/Reaction Time) After a Single Dose of Nasal Spray
Description: Change from baseline in performance on the emotion recognition task (accuracy/reaction time) after a single dose of nasal spray Emotion recognition from point-light displays conveying biological motion.
  Accuracy (acc) is measured in % of correct responses. Reaction time (rt) is measured in milliseconds.
  Higher (accuracy/ reaction time) ratio indicates better performance.
Time Frame: Value at 30 minutes minus value at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in performance (acc/rt ratio)
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 21 | 17
Change in performance (acc/rt ratio) | 0.000029 (0.000069) | 0.000065 (0.000071)

10. Secondary Outcome: Change From Baseline in Performance on the Emotion Recognition Task (Accuracy/ Reaction Time) After 4 Weeks of Nasal Spray
Description: Change from baseline in performance on the emotion recognition task (accuracy/ reaction time) after 4 weeks of nasal spray.
  Emotion recognition from point-light displays conveying biological motion.
  Accuracy (acc) is measured in % of correct responses. Reaction time (rt) is measured in milliseconds.
  Higher (accuracy/ reaction time) ratio indicates better performance.
Time Frame: Value at 4 weeks minus value at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in performance (acc/rt ratio)
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 21 | 17
Change in performance (acc/rt ratio) | 0.000044 (0.000079) | 0.000073 (0.000071)

11. Secondary Outcome: Change From Baseline in Performance on the Emotion Recognition Task (Accuracy/ Reaction Time) After 8 Weeks (Including 4 Weeks Without Nasal Spray)
Description: Change from baseline in performance on the emotion recognition task (accuracy/ reaction time) after 8 weeks (including 4 weeks without nasal spray).
  Emotion recognition from point-light displays conveying biological motion.
  Accuracy (acc) is measured in % of correct responses. Reaction time (rt) is measured in milliseconds.
  Higher (accuracy/ reaction time) ratio indicates better performance.
Time Frame: Value at 8 weeks minus value at baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in performance (acc/rt ratio)
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 21 | 17
Change in performance (acc/rt ratio) | 0.000070 (0.000084) | 0.000088 (0.000089)

12. Secondary Outcome: Change From Baseline in Performance on the Emotion Recognition Task (Accuracy/ Reaction Time) After 52 Weeks (Including 48 Weeks Without Nasal Spray)
Description: Change from baseline in performance on the emotion recognition task (accuracy/ reaction time) after 52 weeks (including 48 weeks without nasal spray)
  Accuracy (acc) is measured in % of correct responses. Reaction time (rt) is measured in milliseconds.
  Higher (accuracy/ reaction time) ratio indicates better performance.
Time Frame: Value at 52 weeks minus value at baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Change in performance (acc/rt ratio)
Groups:
- Syntocinon (Oxytocin, Product Code RVG 03716): Syntocinon (Oxytocin): Syntocinon nasal spray. 4 weeks of a daily single dose (24IU; 3 puffs of 4IU per nostril) of nasal spray
- Placebo (Physiological Water(Sodium Chloride (NaCl) Solution)): Placebo (Physiological water (solution of sodium chloride (NaCl) in water)): Placebo nasal spray.
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 18 | 14
Change in performance (acc/rt ratio) | 0.000071 (0.000079) | 0.000084 (0.000094)

13. Secondary Outcome: Change From Baseline in Informant-based/ Self-report Scores on Questionnaires Assessing Attachment, Social Functioning, Quality of Life and Mood After 4 Weeks of Nasal Spray
Description: The Social Responsiveness Scale (for adults) (SRS-A) uses a four-point Likert-scale. Higher scores indicate lower social responsiveness.
  The Repetitive Behavior Scale - Revised (RBS-R) uses a four-point Likert-scale. Higher scores indicate a higher frequency and/or higher severity of restricted and repetitive behaviors.
  The State Adult Attachment Measure (SAAM) uses a seven-point Likert-scale.Higher scores indicate lower perceived secure attachment on the attachment avoidance and attachment anxiety subscales, and higher perceived secure attachment on the attachment security subscale.
  Inventory of Parent and Peer Attachment (IPPA) uses a four-point Likert-scale. Higher scores indicate indicate increased feelings of secure attachment towards peers or parents.
  World Health Organization Quality of Life - Bref (WHO-QL) uses a five-point Likert scale. Higher scores indicate better quality of life.
  Profile of Mood States (POMS). five-point Likert scale.
Time Frame: Value at 4 weeks minus value at baseline
Population: Intention-to-treat
  Syntocinon:
  IPPA Mother, IPPA Father (n= 21) (listwise missing data: n= 1) SRS-A informant (n= 17) (missing baseline data: n= 5)
  Placebo:
  RBS-R, WHO-QOL (n= 17) (missing baseline data n= 1) SRS-A informant (n= 15) (missing baseline data: n= 3)
Measure: Mean (Standard Deviation); unit: Change from base (units on a scale)
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 22 | 18
Change from base (units on a scale)
  SRS-A self-report | -5.55 (11.40) | -1.06 (10.01)
  SRS-A informant-based: number analyzed (Participants) | 17 | 15
  SRS-A informant-based | 0.0 (15.86) | -0.87 (12.83)
  RBS-R: number analyzed (Participants) | 22 | 17
  RBS-R | -4.77 (6.47) | -1.76 (4.75)
  SAAM avoidance | -0.40 (0.71) | 0.06 (0.98)
  SAAM security | 0.27 (0.77) | 0.05 (0.66)
  SAAM anxiety | -0.14 (0.75) | 0.28 (0.95)
  IPPA Peers | 1.45 (3.85) | 0.56 (4.05)
  IPPA Mother: number analyzed (Participants) | 21 | 18
  IPPA Mother | -0.52 (2.71) | 0.44 (3.45)
  IPPA Father: number analyzed (Participants) | 21 | 18
  IPPA Father | 0.43 (3.30) | -0.61 (3.81)
  WHO-QOL: number analyzed (Participants) | 22 | 17
  WHO-QOL | 1.77 (8.04) | -1.35 (6.74)
  POMS - Tension | -2.00 (2.29) | -2.39 (3.03)
  POMS - Anger | 0.00 (4.05) | -0.61 (2.73)
  POMS - Depression | -1.14 (4.50) | -0.33 (2.81)
  POMS - Vigor | -1.00 (2.53) | -2.94 (3.64)
  POMS - Fatigue | -2.09 (3.99) | -1.11 (5.12)

14. Secondary Outcome: Change From Baseline in Informant-based/ Self-report Scores on Questionnaires Assessing Attachment, Social Functioning, Quality of Life and Mood After 8 Weeks, Including 4 Weeks Without Nasal Spray
Description: as for outcome 13
Time Frame: Value at 8 weeks minus value at baseline
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Change from base (units on a scale)
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 22 | 18
Change from base (units on a scale)
  SRS-A self-report | -5.64 (12.57) | -7.67 (12.09)
  SRS-A informant-based: number analyzed (Participants) | 17 | 15
  SRS-A informant-based | -9.59 (10.98) | -1.20 (10.73)
  RBS-R: number analyzed (Participants) | 22 | 17
  RBS-R | -4.91 (6.33) | -2.35 (3.43)
  SAAM avoidance | -0.38 (0.70) | -0.06 (0.76)
  SAAM security | 0.04 (1.01) | -0.40 (0.99)
  SAAM anxiety | 0.08 (1.05) | 0.11 (0.87)
  IPPA Peers | 1.32 (3.71) | 0.06 (3.70)
  IPPA Mother: number analyzed (Participants) | 21 | 18
  IPPA Mother | -0.38 (3.43) | 0.06 (4.35)
  IPPA Father: number analyzed (Participants) | 21 | 18
  IPPA Father | 0.52 (3.59) | -0.33 (3.87)
  WHO-QOL: number analyzed (Participants) | 22 | 17
  WHO-QOL | 1.14 (5.48) | 0.35 (4.53)
  POMS - Tension | -2.64 (2.80) | -2.11 (3.22)
  POMS - Anger | 0.36 (3.68) | -0.39 (3.91)
  POMS - Depression | -0.82 (2.63) | 0.22 (3.41)
  POMS - Vigor | 0.14 (3.58) | -1.44 (4.33)
  POMS - Fatigue | -2.69 (2.71) | -2.33 (4.47)

15. Secondary Outcome: Change From Baseline in Informant-based/ Self-report Scores on Questionnaires Assessing Attachment, Social Functioning, Quality of Life and Mood After 52 Weeks, Including 48 Weeks Without Nasal Spray
Description: The Social Responsiveness Scale (for adults) (SRS-A) uses a four-point Likert-scale. Higher scores indicate lower social responsiveness.
  The Repetitive Behavior Scale - Revised (RBS-R) uses a four-point Likert-scale. Higher scores indicate a higher frequency and/or higher severity of restricted and repetitive behaviors.
  The State Adult Attachment Measure (SAAM) uses a seven-point Likert-scale.Higher scores indicate lower perceived secure attachment on the attachment avoidance and attachment anxiety subscales, and higher perceived secure attachment on the attachment security subscale.
  Inventory of Parent and Peer Attachment (IPPA) uses a four-point Likert-scale. Higher scores indicate indicate increased feelings of secure attachment towards peers or parents.
  World Health Organization Quality of Life - Bref (WHO-QOL) uses a five-point Likert scale. Higher scores indicate better quality of life.
  Profile of Mood States (POMS). five-point Likert scale.
Time Frame: Value at 52 weeks minus value at baseline
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Change from base (units on a scale)
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 22 | 18
Change from base (units on a scale)
  SRS-A self-report | -8.59 (20.95) | -6.72 (21.01)
  SRS-A informant-based: number analyzed (Participants) | 17 | 15
  SRS-A informant-based | -7.41 (19.26) | -4.13 (24.64)
  RBS-R: number analyzed (Participants) | 22 | 17
  RBS-R | -4.91 (9.46) | -0.41 (4.27)
  SAAM avoidance | -0.52 (1.18) | 0.0 (0.75)
  SAAM security | 0.20 (1.52) | -0.14 (0.66)
  SAAM anxiety | 0.17 (0.94) | 0.11 (1.21)
  IPPA Peers | 0.68 (6.26) | 1.28 (4.17)
  IPPA Mother: number analyzed (Participants) | 21 | 18
  IPPA Mother | 0.33 (3.91) | 1.50 (5.44)
  IPPA Father: number analyzed (Participants) | 21 | 18
  IPPA Father | 0.57 (4.08) | -0.50 (4.53)
  WHO-QOL: number analyzed (Participants) | 22 | 17
  WHO-QOL | 1.14 (8.37) | 0.29 (4.21)
  POMS - Tension | -1.86 (2.29) | -2.28 (3.46)
  POMS - Anger | 0.59 (3.69) | 0.06 (3.84)
  POMS - Depression | 0.50 (2.63) | -0.28 (3.51)
  POMS - Vigor | 1.14 (3.88) | -0.61 (3.27)
  POMS - Fatigue | -0.23 (6.04) | 0.39 (4.73)

16. Secondary Outcome: Change From Baseline in Scores on Questionnaire Assessing Mood After a Single Dose of Nasal Spray
Description: Change from baseline in scores on one questionnaire assessing mood (Profile of Mood States - POMS) after a single dose of nasal spray.
  This instrument comprises emotional adjectives subdivided in five domains: tension (6 items). depression (8 items). vigor (5 items). fatigue (6 items) and anger (7 items) which have to be rated on a five-point Likert scale ranging from 0 (not at all), 1 (a little), 2 (moderately), 3 (quite a lot), to 4 (extremely). Only for the vigor scale, higher scores indicate improvement.
Time Frame: Value at 30 minutes minus value at baseline
Measure: Mean (Standard Deviation); unit: Change from base (units on a scale)
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
Number analyzed (Participants) | 22 | 18
Change from base (units on a scale)
  POMS - Tension | -1.59 (2.11) | -1.39 (2.15)
  POMS - Anger | -0.09 (2.39) | -0.28 (0.89)
  POMS - Depression | -0.23 (1.45) | -0.67 (2.25)
  POMS - Vigor | 0.27 (2.37) | -0.50 (2.38)
  POMS - Fatigue | -1.00 (2.41) | -0.72 (3.68)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of (approximately) four weeks.
Description: Adverse event data were collected via weekly journal entries. In the journal we provided an extensive list of potential adverse events and a blank space below the list to write down adverse events not mentioned in the list. Participants were asked to indicate whether or not they had experienced the event, when it started, how long it lasted, and the severity of the adverse event (mild, moderate, severe).
Arm/Group | Syntocinon (Oxytocin, Product Code RVG 03716) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution))
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 2/22 | 3/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Syntocinon (Oxytocin, Product Code RVG 03716) (N=22) | Placebo (Physiological Water(Sodium Chloride (NaCl) Solution)) (N=18)
Nasal irritation/ runny nose (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) — Nasal irritation/ runny nose due to the nasal spray use

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No